CLINICAL TRIAL: NCT06662721
Title: Baricitinib for Takayasu Arteritis Refractory to TNF-α Inhibitors: a Prospective Pilot Open-label Study
Brief Title: Baricitinib for Refractory Takayasu Arteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liu Tian (Other)
Responsible Party: Sponsor-Investigator, Liu Tian, associate professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU People's Hospital
Record Dates: First submitted 2024-09-18; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Takayasu Arteritis
Keywords: Takayasu arteritis; Baricitinib
MeSH Terms: conditions — Takayasu Arteritis | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Ten patients with Takayasu arteritis refractory to TNF-α inhibitors were treated with baricitinib.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treated with baricitinib (Experimental): Ten patients with Takayasu arteritis refractory TNF-α inhibirors were treated with baricitinib.
  Interventions: Drug: Baricitinib 4 MG

INTERVENTIONS:
Drug: Baricitinib 4 MG — The patients received Baricitinib for 48 weeks. The method is to take Baricitinib 4mg every day for a period of 48 weeks. All the patients will be followed up prospectively for 48 weeks.

SUMMARY:
Takayasu arteritis (TKA) is an autoimmune vasculitis characterized with involvement of aorta and its primary branches. For TKA refractory to TNF-α, Baricitinib, a reversible inhibitor of Janus kinases (JAK) family members JKA1 and JAK2, represents a potential treatment option. This study aims to assess the efficacy and safety of Baricitinib in TKA refractory to TNF-α inhibitors.

DETAILED DESCRIPTION:
This is a multi-center, single-arm trial conducted to evaluate the safety and efficacy of baricitinib in Takayasu arteritis (TKA) refractory to TNF-α inhibitors. Patients in active TKA and unresponsive to at least 6 months of TNF-α inhibitors therapy were enrolled. Patients discontinued TNF-α inhibitors and received baricitinib at 4 mg/day for up to 48 weeks, which was added to the glucocorticoid and immunosuppressants. The clinical manifestations, inflammatory indicators, imaging and treatment of patients were recorded by investigators during the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-70 years at time of screening.
* Diagnosis of Takayasu arteritis (according to the 2022 ACR/EULAR) for ≥3 months before screening.
* Active Takayasu arteritis at time of screening (NIH score≥2).
* Resistant to traditional therapies and anti-TNF-α therapy for at least 12 months.
* Given their written informed consent to participate in the trial and expected to be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* TKA-related active major organ involvement requiring immunosuppressive therapy, e.g., pulmonary (e.g., pulmonary artery aneurysm), vascular (e.g., thrombophlebitis, recurrent malignant aneurysms), gastrointestinal (e.g., gastrointestinal ulcers), and central nervous system (e.g., meningoencephalitis).
* High-dose glucocorticoid (>1mg/kg/d) usage within 1 month.
* Severe comorbidities: including heart failure (≥ grade III NYHA), renal insufficiency (creatinine clearance ≤30 ml/min), hepatic insufficiency (serum ALT or AST >3 times the ULN, or total bilirubin >ULN for the central laboratory conducting the test). Other severe, progressive or uncontrolled hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis).
* Known allergies, hypersensitivity, or intolerance to Baricitinib or its excipients.
* Had a severe infection (including, but not limited to hepatitis, pneumonia, sepsis, or pyelonephritis); had been hospitalized for an infection; or had been treated with IV antibiotics for an infection, within 2 months prior to the first administration of study agent.
* Chest radiograph within 3 months prior to the first administration of study agent that showed an abnormality suggestive of a malignancy or current active infection, including tuberculosis.
* Infected with HIV (positive serology for HIV antibody) or hepatitis C (positive serology for Hep C antibody). If seropositive, consultation with a physician with expertise in the treatment of HIV or hepatitis C virus infection was recommended.
* Infected with hepatitis B virus. For patients who were not eligible for this study due to hepatitis B virus test results, consultation with a physician with expertise in the treatment of hepatitis B virus infection was recommended.
* Had any known malignancy or has a history of malignancy within the previous 5 years (with the exception of a nonmelanoma skin cancer that had been treated with no evidence of recurrence for ≥3 months before the first study agent administration or cervical neoplasia with surgical cure).
* Had uncontrolled psychiatric or emotional disorder, including a history of drug and alcohol abuse within the past 3 years that might prevent the successful completion of the study.
* Received, or was expected to receive, any live virus or bacterial vaccination within 3 months before the first administration of study agent, during the study, or within 4 months after the last administration of study agent. Had a BCG vaccination within 12 months of screening.
* Pregnancy, lactation or women of child-bearing potential (WCBP) unwilling to use medically approved contraception whilst receiving treatment and for 12 months after treatment has finished.
* Men whose partners are of child-bearing potential but who are unwilling to use appropriate medically approved contraception whilst receiving treatment and for 12 months after treatment has finished.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Patients achieving complete remission and partial remission | Week 24
  The primary endpoint was defined as the proportion(percent) of patients in the whole cohort achieving complete remission and partial remission by week 24.

SECONDARY OUTCOMES:
Changes of National Institutes of Health (NIH) score of patients | Week 24 and week 48
  The manifestations, imaging findings and laboratory parametes were recorded during the follow-up. The disease activity of patients were accessed by National Institutes of Health (NIH) score. (Range: 0~4, higher scores mean higher disease activity)
Changes of Indian Takayasu Clinical Activity Score (ITAS2010) of patients | Week 24 and week 48
  The manifestations, imaging findings and laboratory parameters were recorded during the follow-up. The disease activity of patients were accessed by Indian Takayasu Clinical Activity Score (ITAS2010). (Range: 0~51, higher scores mean higher disease activity)
Changes of C-reactive protein | Week 24 and week 48
  Blood samples were collected from all patients and the concentration of C-reactive protein (mg/L) were recorded.
Changes of erythrocyte sedimentation rate | Week 24 and week 48
  Blood samples were collected from all patients and the erythrocyte sedimentation rates (mm/h) were recorded.
Changes of dosage of glucocorticoids from baseline. | Week 24 and week 48
  The dosage of glucocorticoids (mg/day) of all patients were recorded during the follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li J, Xia W, Ji H, Gong X, Dong Q, Wu Y, Wang L, Peng M, Liu J, Ma K, Yu Q, Cui X, Luo Y, Zhu W, Zhang S, Chen S, Li Y, Li Z, Liu T. Baricitinib for Takayasu arteritis refractory to TNF-alpha inhibitors: a multicentre, single-arm trial. Rheumatology (Oxford). 2025 Oct 1;64(10):5262-5268. doi: 10.1093/rheumatology/keaf286. PMID 40411764